CLINICAL TRIAL: NCT02383485
Title: Exercise and Overweight Children's Cognition (Supplement)
Brief Title: Nonalcoholic Fatty Liver Disease and Atherosclerotic Risk in Children
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Catherine Davis, Professor of Pediatrics, Graduate Studies and Physiology, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HL087923-02S1 (NIH); R01HL087923-02S1 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Overweight and Obesity; Non-alcoholic Fatty Liver Disease
Keywords: arterial stiffness
MeSH Terms: conditions — Overweight; Obesity; Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- After-school exercise program (Experimental): 40 min/day vigorous aerobic games after school
  Interventions: Behavioral: Exercise; Behavioral: After-school program
- Sedentary after-school program (Active Comparator): Attention-control condition similar to experimental condition with the exception of exercise
  Interventions: Behavioral: After-school program

INTERVENTIONS:
Behavioral: Exercise — Heart rate monitors worn by each child at each session
  Other Names: Aerobic training
  Arms: After-school exercise program
Behavioral: After-school program — Supervised recreational program with token economy

SUMMARY:
Nonalcoholic fatty liver disease is a serious health condition in overweight children which can lead to heart disease. This project will examine the links between liver health and cardiovascular risk factors in overweight and obese children, and will test the effect of a long-term after-school exercise program.

Provision of comprehensive evidence for the benefits of exercise on children's health may reduce barriers to vigorous physical activity programs during a childhood obesity epidemic.

DETAILED DESCRIPTION:
This is an ancillary study adding cardiometabolic outcome measures to an ongoing NIH-funded randomized trial of exercise in overweight children ("SMART study," R01 HL087923, P.I. Davis, NCT02227095). This presents the opportunity to obtain detailed measures of liver and vascular health to provide information about the effects of exercise on these conditions.

ELIGIBILITY:
Inclusion Criteria:

* 8-11 years of age
* Overweight or obese (BMI-for-age >= 85th percentile)
* Able to participate in exercise testing and intervention
* Participating in the SMART Study

Exclusion Criteria:

* Medical condition or medications that would interfere with measurements
* Participation in weight control or formal exercise program outside physical education that meets more than 1 day/week
* T-score > 75 on the BRIEF Behavior Regulation scale to avoid program disruption
* Unable to complete magnetic resonance imaging.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2008-05; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Liver Fat | Baseline, 8 Months
  Change in the proportion of liver fat via MRI
Change in Arterial Stiffness | Baseline, 8 Months
  Change in carotid-femoral pulse wave velocity

SECONDARY OUTCOMES:
Change in Liver Fibrosis | Baseline, 8 Months
  Change in Fibroscan transient elastography measure
Change in Liver Inflammation | Baseline, 8 Months
  Change in ratio of aspartate aminotransferase to alanine aminotransferase (AST/ALT), C-reactive protein
Change in Quality of Life | Baseline, 8 Months
  Change in PedsQL questionnaire responses
Associations among Liver Fat, Fibrosis and Inflammation, Arterial Stiffness, and Other Cardiovascular Risk Indices | Baseline
  At baseline, the proportion of liver fat (ascertained by MRI) will be closely related to indices of liver fibrosis (as detected by transient elastography) and inflammation (ratio of aspartate aminotransferase to alanine aminotransferase, AST/ALT; C-reactive protein, CRP), and to arterial stiffness and other indices of cardiovascular risk (body fat (DXA), visceral fat (MRI), aerobic fitness, insulin resistance, adiponectin, dyslipidemia).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Davis, PhD, Principal Investigator — 706-721-9551
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States